CLINICAL TRIAL: NCT05820776
Title: Remote Exercise-based Pulmonary Rehabilitation Telemedicine in Chronic Respiratory Disease: an Observational Cohort Study
Brief Title: Tele-rehabilitation in Chronic Respiratory Disease: an Observational Cohort Study
Status: Recruiting | Type: Observational
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Director, Program in Respiratory Rehabilitation, West Park Healthcare Centre
Other Study IDs: PTR-RG2023
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Chronic Respiratory Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pulmonary rehabilitation — The intervention is PR delivered via a telemedicine. The intervention is PR delivered via a telemedicine. The program is delivered by the multidisciplinary via a remote application for two sessions per week for ten weeks. Remotely supervised exercise includes: 1) deep breathing reinforcing pursed lip and diaphragmatic breathing; 2) warm up breathing and stretching exercise; 3) a cardiorespiratory aerobic exercise battery; 4) resistance training, and; stretching cool down. There is also an educational component. The secondary (maintenance) program includes ongoing remotely supervised exercise and education once a week for six months (24 sessions). All patients successfully completing the initial PR are offered the maintenance program.

SUMMARY:
Pulmonary rehabilitation is a program that helps people with lung disease improve their function. It uses exercise, education, and self-management strategies to improve physical ability and quality of life. Because some people are unable to visit West Park Healthcare Centre, we established a remote supervised pulmonary rehabilitation program that patients can access via an electronic device (computer, tablet or smart phone). Regular quality assurance is necessary to ensure that the program is effective. We plan to collect and summarize the program's results. The benefit of doing so is that it allows us to make any changes or improvements that may help patients with chronic respiratory conditions.

ELIGIBILITY:
Inclusion Criteria:

* stable chronic respiratory disease
* qualified candidates for pulmonary rehabilitation,
* current non-smoker;
* primary diagnosis chronic respiratory disease limited by dyspnea (mMRC≥2);
* free of exacerbation at the time of admission, and
* stable co-existing conditions

Exclusion Criteria:

* completed PR within the previous 12 months of the current admission and
* being unable to communicate with the treating team.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with chronic respiratory disease affecting the airways and other structures of the lungs causing dyspnea including chronic obstructive pulmonary disease (COPD), occupational lung diseases and pulmonary hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
health-related quality of life Chronic Respiratory Questionnaire - dyspnea | 12 weeks
  Disease-specific health-related quality of life questionnaire. Developed to measure the impact of Chronic Obstructive Pulmonary Disease (COPD) on a person's life.

SECONDARY OUTCOMES:
6-minute walk test distance | 12 weeks
  An objective evaluation of functional exercise capacity; the subject is asked to walk as far as possible for 6 minutes.
30-second Chair Stand Test | 12 weeks
  A measurement to assess functional leg strength and endurance by involves recording the number of stands a person can complete in 30 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Roger Goldstein, MD, Principal Investigator — West Park Healthcare Centre
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No